CLINICAL TRIAL: NCT02918825
Title: A Randomized Trial to Compare the Efficiency and Side Effect Between Olanzapine and Long-acting Paliperidone Palmitate Injection in Schizophrenia
Brief Title: Long-acting Paliperidone Palmitate Injection and Olanzapine for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Director of Biological psychiatry center,, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WZKN-sch
Record Dates: First submitted 2016-09-20; First posted 2016-09-29 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; clinical trial; olanzapine; paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paliperidone (Experimental): Drug: Paliperidone, 75-150mg/month, once a month, 12 weeks
  Interventions: Drug: Paliperidone
- Olanzapine (Active Comparator): Drug: Olanzapine, 20mg/day, twice a day, 12 weeks
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine
  Arms: Olanzapine
Drug: Paliperidone — Paliperidone
  Arms: Paliperidone

SUMMARY:
A randomized trial of olanzapine and Long-acting paliperidone palmitate injection in the treatment of 100 treatment- naive first-episode patients with schizophrenia.

DETAILED DESCRIPTION:
OBJECTIVE: Investigator compared the efficiency, social function, cognitive function and side effect of olanzapine and Long-acting paliperidone palmitate injection in the treatment of first-episode drug-naive patients with schizophrenia.

METHODS:

1. Clinical Trial: This is a randomized trial in treatment-naive first-episode patients with schizophrenia. The study consists of a 1-week stabilization phase, followed by 12 weeks of treatment. The total trial duration is 13 weeks.
2. Assessment Procedures:

2.1. Primary Outcome Variable-psychopathology: Assessment instruments include the Positive and Negative Syndrome Scale (PANSS), the Assessment of Negative Symptoms (SANS) and the Clinical Global Impression (ICG). Patients are interviewed at screening, at week-4, at week-1, at baseline and at every two weeks, for a total of 12 ratings.

2.2. Cognitive tests: A comprehensive battery of tests encompassing the cognitive domains of executive function, attention, memory, perception, and general intellect is administered twice at baseline and at the end of 16-week treatment by a trained psychologist. Scoring follows standardized procedures. The Wisconsin Card Sorting Test (WCST) is administered as a measure of executive function. The N-back (0-3 back) test is administered as a measure of working memory. Logical Memory I and II, Verbal Paired Associates I and II, Visual Reproduction I and II and Digits Forward from the Wechsler Memory Scale-Revised (WMS-R) are administered as a tests of episodic memory. The Distractibility version of Gordon Continuous Performance Test (CPT)is administered as a test of attention. A four-subtest version of the Wechsler Adult Intelligence Scale-Revised (WAIS-R), consisting of the Arithmetic, Similarities, Picture Completion, and Digit Symbol Substitution tests is administered to obtain an estimate of current Full- Scale Intelligence Quotient (FSIQ).

2.3. Social functioning: The Personal and Social Performance Scale (PSP) examines the four dimensions of social functioning: Socially useful activities including work and study, personal and social relationships, self-care, disturbing and aggressive behaviors.

2.4. Side Effects: Parkinsonism is rated with the Simpson-Angus Scale for extrapyramidal side effects (SAS). The Abnormal Involuntary Movement Scale (AIMS) is chosen to assess tardive dyskinesia (TD) severity. All of the AIMS and Simpson-Angus Rating Scales are administered by the same investigator, at screening, at week-4, at week-1, at baseline and at baseline and at every two weeks, for a total of 12 ratings.

2.5.Weight gain measurement: weight gain every week 2.6. Serum measurement: triglyceride, blood sugar，cholesterol，blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizophreniform disorder;
* Duration of symptoms not longer than 60 months;
* No prior treatment with antipsychotic medication or, if previously treated, a total lifetime usage of less than 14 days;
* Between 18 and 45 years of age; and
* Current psychotic symptoms of moderate severity.

Exclusion Criteria:

* A DSM-IV Axis I diagnosis other than schizophrenia or schizophreniform;
* Documented disease of the central nervous system that can interfere with the trial assessments including, but not limited to stroke, tumor, Parkinson's disease, Huntington's disease, seizure disorder, history of brain trauma resulting in significant impairment, chronic, infection;
* Acute, unstable and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension);
* A clinically significant ECG abnormality in the opinion of the investigator;
* Pregnant or breast-feeding female;
* Use of disallowed concomitant therapy;
* History of severe allergy or hypersensitivity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Symptoms assessed on PANSS. | 12 weeks
  Clinical symptoms

SECONDARY OUTCOMES:
Clinical global impression assessed on CGI. | 12 weeks
  clinical severity
Cognitive functioning assessed on RBANS. | 12 weeks
  cognitive performance
Number of weight change in treatment assessed on Weight gain. | 12 weeks
  weight gain
Abnormal Involuntary Movement Scale assessed Abnormal Involuntary Movement Scale assessed on AIMS. | 12 weeks
  Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhang, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data will be available on request

REFERENCES:
- [Result] Kim E, Correll CU, Mao L, Starr HL, Alphs L. Once-monthly paliperidone palmitate compared with conventional and atypical daily oral antipsychotic treatment in patients with schizophrenia. CNS Spectr. 2016 Dec;21(6):466-477. doi: 10.1017/S1092852916000444. Epub 2016 Sep 15. PMID 27629292
- [Result] Yoshimura R, Hori H, Katsuki A, Atake K. Marked Improvement of Meige Syndrome in a Japanese Male Patient with Schizophrenia After Switching from Risperidone to Paliperidone: A Case Report. J UOEH. 2016 Sep;38(3):233-6. doi: 10.7888/juoeh.38.233. PMID 27627971
- [Result] Young-Xu Y, Duh MS, Muser E, DerSarkissian M, Faust E, Kageleiry A, Bhak RH, Fu DJ, Lefebvre P, Shiner B. Impact of Paliperidone Palmitate Versus Oral Atypical Antipsychotics on Health Care Resource Use and Costs in Veterans with Schizophrenia. J Clin Psychiatry. 2016 Oct;77(10):e1332-e1341. doi: 10.4088/JCP.16m10745. PMID 27574835